CLINICAL TRIAL: NCT06938646
Title: Microbiome Characterization in Patients With Fatty Pancreas: a Pilot Cohort Study
Brief Title: Microbiome Characterization in Fatty Pancreas
Acronym: FPM1
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2024.585
Record Dates: First submitted 2025-04-08; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Fatty Pancreas; Microbiome Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Stool sample
  One bottle of stool specimen will be collected in sterile container. The collected stool specimen will be placed on ice and promptly transferred to a -80°C refrigerator for cryopreservation.
  Blood sample
  10ml of blood will be collected in ethylenediaminetetraacetic acid (EDTA) tubes. The collected blood sample will be promptly transferred to a -80°C refrigerator for cryopreservation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with fatty pancreas: Patients who underwent MRI-PDFF for pancreatic fat fraction and liver fat fraction measurements between 1/2022 and 11/2024 for evaluation of FP and fatty liver in GI and hepatology clinics of the Prince of Wales Hospital will be screened for eligibility of this study. Each patient with FP will be matched by sex and age (+/- 3 years) with 1 patient without FP (MRI-PDFF pancreatic fat fraction < 6.2%). Patients with significant alcohol consumption, defined as alcohol intake of over 20g daily (140g weekly) for men and 10g daily (70g weekly) for women will be excluded.
- Healthy subjects: Healthy subjects

SUMMARY:
There has been a growing interest in evaluating the role of gut and intra-lesional microbiome in the pathogenesis of various benign and malignant conditions of the GI tract, liver and pancreas. In addition, the feasibility of using microbiome signature as non-invasive biomarker for benign and malignant disease conditions of the GI tract has also been studied. While research on the impact of microbiome and genomics has been conducted in some pancreatic disorders such as acute pancreatitis, pre-malignant mucinous pancreatic cystic neoplasms (eg, IPMN) and pancreatic cancer, very little data is available regarding the microbiome signature and genomics associated with FP. As such, it would be clinically important to conduct a pilot study to investigate the microbiome and genomics associated in patients with or without FP defined by MRI-PDFF pancreatic fat fraction measurement.

DETAILED DESCRIPTION:
Fatty pancreas (FP) is a pathological metabolic condition characterized by excessive intra-pancreatic fat deposition (IPFD). FP is an increasingly recognized metabolic condition with a prevalence of 16% to 35% in Asian populations. While ultrasound, computed tomography (CT) and magnetic resonance imaging (MRI) have been used for fat quantitation in organs, MRI is best suited for this purpose since its signal is dependent on fat content. Quantitative proton density fat fraction measurement by MRI (MRI-PDFF) is regarded as the current gold standard for fat quantification in organs such as liver and pancreas since the fat fraction measurements by MRI are reproducible, accurate and have been validated against histology. In a meta-analysis of 9 studies using MRI for pancreatic fat quantification, the upper limit of normal of pancreatic fat in healthy subjects was 6.2%.

FP has gained clinical attention since FP has been associated with both benign and malignant diseases of the pancreas. For example, recent retrospective studies have suggested an increased risk of pancreatic cancer, intraductal papillary mucinous neoplasms (IPMN) and neoplastic progression of Branch Duct type IPMN (BD-IPMN) in patients with FP defined by computed tomography (CT) attenuation indexes . In another retrospective study of 62 patients using MRI-PDFF for pancreatic fat quantification, high pancreatic fat fraction was associated with high-risk IPMN in surgical specimen. In a community cohort study of 685 adult Chinese volunteers, our team was the first to report on the prevalence of FP (16.1%) in Hong Kong adults using MRI for pancreatic fat quantification in 2014 . In our recently published 10-year prospective follow-up study of the same cohort, FP was independently associated with subsequent diabetes development.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients with FP, defined by MRI-PDFF pancreatic fat fraction > 6.2%
* Patients who are able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Unable to provide written informed consent
* Recent use of antibiotic, prebiotic, probiotic and symbiotic
* Patients with significant alcohol consumption, defined as alcohol intake of over 20 g daily (140 g weekly) for men and 10 g daily (70 g weekly) for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent MRI-PDFF for pancreatic fat fraction and liver fat fraction measurements between 1/2022 and 11/2024 for evaluation of FP and fatty liver in GI and hepatology clinics of the Prince of Wales Hospital will be screened for eligibility of this study. Each patient with FP will be matched by sex and age (+/- 3 years) with 1 patient without FP (MRI-PDFF pancreatic fat fraction < 6.2%). Patients with significant alcohol consumption, defined as alcohol intake of over 20g daily (140g weekly) for men and 10g daily (70g weekly) for women will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome in patients with FP | At the time of procedure
  Characterization of the gut microbiome in patients with FP (defined by MRI-PDFF pancreatic fat fraction > 6.2%) and age-sex matched subjects without FP

SECONDARY OUTCOMES:
Gut microbiome in patients with FP and co-existing fatty liver, patients with FP alone, patients with fatty liver alone, and patients without FP and fatty liver | At the time of procedure
  To evaluate the difference in gut microbiome in patients with FP and co-existing fatty liver (defined by MRI-PDFF intrahepatic fat fraction > 5%), patients with FP alone, patients with fatty liver alone, and patients without FP and fatty liver
Correlation of gut microbiome in the subgroup of patients with FP and mucinous pancreatic cystic size and presence of worrisome features | At the time of procedure
  To correlate the gut microbiome in the subgroup of patients with FP and mucinous pancreatic cystic neoplasms (PCN) (eg, IPMN) with PCN size and presence of worrisome features defined by the 2024 Kyoto evidence-based consensus guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No